CLINICAL TRIAL: NCT03578809
Title: A Randomized, Placebo-controlled Phase 2b Study to Evaluate the Safety and Efficacy of MEDI6012 in Acute ST Elevation Myocardial Infarction
Brief Title: A Study to Evaluate the Safety and Efficacy of MEDI6012 in Acute ST Elevation Myocardial Infarction
Acronym: REAL-TIMI 63B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: The TIMI Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5780C00007
Record Dates: First submitted 2018-06-08; First posted 2018-07-06 (Actual); Results first posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: In this study, the participant and sponsor staff will be blinded. Sites will be trained to keep the investigator blinded. However, due to the acute nature of the study, members of the research team and, possibly, the investigator may be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort A: Placebo (Placebo Comparator): Participants will receive placebo matched to MEDI6012 on Day 1 prior to pPCI followed by a second inpatient dose on Day 3 by IV push.
  Interventions: Other: Placebo
- Cohort A: MEDI6012 (Experimental): Participants will receive loading dose of MEDI6012 300 mg on Day 1 prior to pPCI followed by a second inpatient dose of MEDI6012 150 mg on Day 3 by IV push.
  Interventions: Biological: MEDI6012
- Cohort B: Placebo (Placebo Comparator): Participants will receive placebo matched to MEDI6012 on Day 1 prior to pPCI followed by a second inpatient dose on Day 3, and outpatient maintenance doses on Days 10, 17, 24, and 31 by IV push.
  Interventions: Other: Placebo
- Cohort B: MEDI6012 (Experimental): Participants will receive loading dose of MEDI6012 300 mg on Day 1 prior to pPCI followed by a second inpatient dose of MEDI6012 150 mg on Day 3, and outpatient maintenance doses of MEDI6012 100 mg on Days 10, 17, 24, and 31 by IV push.
  Interventions: Biological: MEDI6012

INTERVENTIONS:
Biological: MEDI6012 — MEDI6012
  Other Names: MEDI6012 300 mg will be administered on Day 1 and MEDI6012 150 mg on Day 3 by IV push in Cohorts A and B. In Cohort B, MEDI6012 100 mg will be administered on Days 10, 17, 24, and 31 by IV push.
  Arms: Cohort A: MEDI6012; Cohort B: MEDI6012
Other: Placebo — Placebo
  Other Names: Placebo matched to MEDI6012 will be administered on Day 1 and Day 3 by IV push in Cohorts A and B, and on Days 10, 17, 24, and 31 by IV push in Cohort B.
  Arms: Cohort A: Placebo; Cohort B: Placebo

SUMMARY:
This is a Phase 2b randomized, blinded, placebo controlled study to evaluate the efficacy, safety, PK/pharmacodynamic, and immunogenicity of repeat doses of MEDI6012 in adult participants presenting with acute STEMI (ST segment elevation myocardial infarction).

The study will enrol participants presenting with acute STEMI who are planned for primary percutaneous coronary intervention (pPCI). For all participants, an end of study CMR will be performed at 10-12 weeks (70-84 days following Dose 1). A subset of participants will also undergo an index and an end of study CTA.

ELIGIBILITY:
Inclusion Criteria:

* Acute STEMI (ST segment elevation myocardial infarction) diagnosed by ST elevation
* Planned for primary PCI (percutaneous coronary intervention)
* Men and women without child-bearing potential aged 30-80 years of age
* Capable and willing to provide informed consent.
* Capable of completing study visits

Exclusion Criteria:

* Fibrinolytic administration for index event
* Known prior MI or prior coronary artery bypass graft (CABG) surgery
* Known pre-existing cardiomyopathy
* History of anaphylaxis
* Suspected non-thrombotic etiology (ie, vasospasm, dissection, Takotsubo cardiomyopathy)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 593 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- Brazil (3):
  - Research Site, Belo Horizonte
  - Research Site, Campinas
  - Research Site, Porto Alegre
- Czechia (6):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Liberec
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Ústí nad Labem
- Research Site, Budapest, Hungary
- Israel (6):
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Netherlands (2):
  - Research Site, Alkmaar
  - Research Site, Nijmegen
- Poland (2):
  - Research Site, Bydgoszcz
  - Research Site, Lodz
- Russia (2):
  - Research Site, Kazan'
  - Research Site, Saint Petersburg
- Slovakia (2):
  - Research Site, Banská Bystrica
  - Research Site, Nitra
- Spain (2):
  - Research Site, Madrid
  - Research Site, Pontevedra
- United Kingdom (3):
  - Research Site, Dundee
  - Research Site, Leeds
  - Research Site, Stevenage

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Bonaca MP, Morrow DA, Bergmark BA, Berg DD, Lima JAC, Hoffmann U, Kato Y, Lu MT, Kuder J, Murphy SA, Spinar J, Oude Ophuis T, Kiss RG, Lopez-Sendon J, Averkov O, Wheatcroft SB, Kubica J, Carlos Nicolau J, Furtado RHM, Abuhatzira L, Hirshberg B, Omar SA, Vavere AL, Chang YT, George RT, Sabatine MS. Randomized, Placebo-Controlled Phase 2b Study to Evaluate the Safety and Efficacy of Recombinant Human Lecithin Cholesterol Acyltransferase in Acute ST-Segment-Elevation Myocardial Infarction: Results of REAL-TIMI 63B. Circulation. 2022 Sep 20;146(12):907-916. doi: 10.1161/CIRCULATIONAHA.122.059325. Epub 2022 Aug 30. PMID 36039762
- See also: D5780C00007 CSP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5780C00007&attachmentIdentifier=f9c1bc23-394a-4215-977e-3838819a18ee&fileName=d5780c00007-csp-amendment-6_redacted_Final_Redacted.pdf&versionIdentifier=
- See also: D5780C00007 SAP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5780C00007&attachmentIdentifier=526e518e-a4f4-4233-a41b-438cf3d63bb1&fileName=d5780c00007-16-1-9-statistical-analysis-plan-v3.0_redacted_final_Redacted.pdf&versionIdentifier=
- See also: D5780C00007 CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5780C00007&attachmentIdentifier=c59933fe-bdf0-49d6-b9f6-5e903e19d07b&fileName=d5780c00007-study-synopsis_redacted_final_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 10 countries (Brazil, Czech Republic, Hungary, Israel, Netherlands, Poland, Russian Federation, Slovakia, Spain, and the United Kingdom).
Pre-assignment Details: In total, 593 participants were randomized into the study and 575 participants were treated with the study drug.
Groups:
- Cohort A: Placebo: Participants received placebo matched to MEDI6012 on Day 1 prior to primary percutaneous coronary intervention (pPCI) followed by a second inpatient dose on Day 3 by intravenous (IV) push.
- Cohort A: MEDI6012: Participants received loading dose of MEDI6012 300 mg on Day 1 prior to pPCI followed by a second inpatient dose of MEDI6012 150 mg on Day 3 by IV push.
- Cohort B: Placebo: Participants received placebo matched to MEDI6012 on Day 1 prior to pPCI followed by a second inpatient dose on Day 3, and outpatient maintenance doses on Days 10, 17, 24, and 31 by IV push.
- Cohort B: MEDI6012: Participants received loading dose of MEDI6012 300 mg on Day 1 prior to pPCI followed by a second inpatient dose of MEDI6012 150 mg on Day 3, and outpatient maintenance doses of MEDI6012 100 mg on Days 10, 17, 24, and 31 by IV push.
Period: Overall Study
Arm/Group | Cohort A: Placebo | Cohort A: MEDI6012 | Cohort B: Placebo | Cohort B: MEDI6012
Started | 94 | 185 | 112 | 202
Treated | 90 | 179 | 111 | 195
Completed | 88 | 171 | 108 | 193
Not Completed | 6 | 14 | 4 | 9
Not completed — Death | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 5 | 2 | 0
Not completed — Other | 3 | 6 | 2 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants, grouped according to assigned treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Placebo | Cohort A: MEDI6012 | Cohort B: Placebo | Cohort B: MEDI6012 | Total
Number analyzed (Participants) | 94 | 185 | 112 | 202 | 593
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.7 (10.3) | 59.9 (10.2) | 62.6 (10.8) | 59.9 (10.0) | 60.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 35 | 27 | 49 | 131
  Male | 74 | 150 | 85 | 153 | 462
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 8 | 2 | 10 | 22
  Not Hispanic or Latino | 92 | 177 | 110 | 192 | 571
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 2 | 3
  White | 94 | 182 | 110 | 194 | 580
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Global Infarct Size
Description: Global infarct size expressed as a percentage of left ventricle (LV) mass measured on delayed-enhanced cardiovascular magnetic resonance (CMR) imaging in 10-12 weeks post myocardial infarction (MI) is reported.
Time Frame: 70 to 84 days post Day 1 dose
Population: Primary efficacy analysis population included randomized participants with a Thrombolysis in Myocardial Infarction (TIMI) flow Grade 0-1 on initial angiography who received at least 2 doses of study drug and grouped according to assigned treatment. 'Number of participants analyzed' denotes the number of participants evaluated for this outcome measure.
Measure: Geometric Mean (90% Confidence Interval); unit: Percentage of global infarct size
Arm/Group | Cohort A: Placebo | Cohort A: MEDI6012 | Cohort B: Placebo | Cohort B: MEDI6012
Number analyzed (Participants) | 43 | 97 | 61 | 108
Percentage of global infarct size | 5.453 [3.781 to 7.865] | 8.598 [7.228 to 10.229] | 9.004 [7.219 to 11.230] | 7.819 [6.658 to 9.183]

2. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: The LVEF measured by cine magnetic resonance imaging (MRI) at 10-12 weeks post-MI is reported.
Time Frame: 70 to 84 days post Day 1 dose
Population: Primary efficacy analysis population included randomized participants with a TIMI flow Grade 0-1 on initial angiography who received at least 2 doses of study drug and grouped according to assigned treatment. 'Number of participants analyzed' denotes the number of participants evaluated for this outcome measure.
Measure: Geometric Mean (90% Confidence Interval); unit: Percentage of LVEF
Arm/Group | Cohort A: Placebo | Cohort A: MEDI6012 | Cohort B: Placebo | Cohort B: MEDI6012
Number analyzed (Participants) | 43 | 99 | 61 | 108
Percentage of LVEF | 47.626 [44.344 to 51.152] | 47.083 [45.167 to 49.079] | 47.329 [45.158 to 49.604] | 49.722 [48.117 to 51.381]

3. Secondary Outcome: Change in Non-calcified Plaque Volume (NCPV) in the Coronary Arteries in Cohort B
Description: Change in NCPV in the coronary arteries from index computed tomography angiography (CTA) to 10-12 weeks post-MI is reported. The index CTA was preferably to be performed between 48 to 72 hours post Dose 1 (could be done up to 5 days post Dose 1) but no earlier than 40 hours post Dose 1. Participants with creatinine clearance >= 60 mL/min (Cockcroft Gault equation) within 6 hours underwent an index coronary CTA no earlier than 40 hours following the first dose.
Time Frame: Day 1 dose (48 to 72 hours post Dose 1) through 70 to 84 days post Day 1 dose
Population: The CTA analysis population included randomized participants in the 6-dose regimen who received a full treatment course of study drug, were eligible, and had coronary CTA. 'Number of participants analyzed' denotes the number of participants evaluated for this outcome measure.
Measure: Geometric Mean (90% Confidence Interval); unit: mm^3
Arm/Group | Cohort B: Placebo | Cohort B: MEDI6012
Number analyzed (Participants) | 60 | 121
mm^3 | 1.049 [0.915 to 1.203] | 0.998 [0.919 to 1.085]

4. Secondary Outcome: Left Ventricular Mass by Late Gadolinium Enhancement (LGE)
Description: The left ventricular mass by LGE is reported.
Time Frame: 70 to 84 days post Day 1 dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Cohort A: Placebo | Cohort A: MEDI6012 | Cohort B: Placebo | Cohort B: MEDI6012
Number analyzed (Participants) | 43 | 97 | 61 | 108
g | 119.740 (31.384) | 119.581 (23.949) | 115.221 (28.328) | 117.920 (24.821)

5. Secondary Outcome: Left Ventricular Mass by Cine Magnetic Resonance Imaging (MRI)
Description: The left ventricular mass by cine MRI is reported.
Time Frame: 70 to 84 days post Day 1 dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Cohort A: Placebo | Cohort A: MEDI6012 | Cohort B: Placebo | Cohort B: MEDI6012
Number analyzed (Participants) | 43 | 99 | 61 | 108
g | 113.953 (31.261) | 113.870 (23.885) | 110.244 (28.009) | 111.533 (23.329)

6. Secondary Outcome: Left Ventricular End-diastolic and End-systolic Volume
Description: Left ventricular end-diastolic and end-systolic volume is reported.
Time Frame: 70 to 84 days post Day 1 dose
Population: as for outcome 2
Measure: Geometric Mean (90% Confidence Interval); unit: mL
Arm/Group | Cohort A: Placebo | Cohort A: MEDI6012 | Cohort B: Placebo | Cohort B: MEDI6012
Number analyzed (Participants) | 43 | 99 | 61 | 108
mL
  Left ventricular end-diastolic volume | 174.059 [161.956 to 187.066] | 176.523 [169.259 to 184.098] | 167.480 [157.010 to 178.649] | 172.733 [166.031 to 179.706]
  Left ventricular end-systolic volume | 87.038 [78.229 to 96.838] | 89.594 [83.818 to 95.768] | 84.977 [77.205 to 93.532] | 83.676 [78.606 to 89.073]

7. Secondary Outcome: Left Ventricular End-diastolic and End-systolic Volume Index
Description: Left ventricular end-diastolic and end-systolic volume index is reported.
Time Frame: 70 to 84 days post Day 1 dose
Population: as for outcome 2
Measure: Geometric Mean (90% Confidence Interval); unit: mL/m^2
Arm/Group | Cohort A: Placebo | Cohort A: MEDI6012 | Cohort B: Placebo | Cohort B: MEDI6012
Number analyzed (Participants) | 42 | 99 | 61 | 108
mL/m^2
  Left ventricular end-diastolic volume index | 89.158 [84.324 to 94.269] | 90.280 [86.818 to 93.880] | 86.118 [81.401 to 91.107] | 87.258 [84.211 to 90.416]
  Left ventricular end-systolic volume index | 44.491 [40.537 to 48.830] | 45.821 [42.970 to 48.863] | 43.695 [40.024 to 47.703] | 42.270 [39.845 to 44.842]

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through Day 195 post Day 1 dose
Population: As-treated population included all treated participants, grouped according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo | Cohort A: MEDI6012 | Cohort B: Placebo | Cohort B: MEDI6012
Number analyzed (Participants) | 90 | 179 | 111 | 195
Participants
  Any TEAEs | 49 | 114 | 70 | 136
  Any TESAEs | 11 | 34 | 24 | 41

9. Secondary Outcome: Serum Concentration of MEDI6012 (Lecithin-cholesterol Acyltransferaes [LCAT] Mass)
Description: Serum concentration of MEDI6012 is reported.
Time Frame: Pre- and post-dose on Days 1, 3, 17, and 31
Population: Pharmacokinetic population included all participants in the As-treated population who had at least one detectable serum concentration measurement for LCAT mass or activity. 'Number analyzed' denotes participants who had adequate pharmacokinetic sample of MEDI6012 for the specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A: MEDI6012 | Cohort B: MEDI6012
Number analyzed (Participants) | 179 | 193
ng/mL
  Day 1 (pre-dose): number analyzed (Participants) | 3 | 6
  Day 1 (pre-dose) | NA (NA) — Data were not calculated because the concentration was below limit of quantification. | NA (NA) — Data were not calculated because the concentration was below limit of quantification.
  Day 1 (post-dose): number analyzed (Participants) | 172 | 183
  Day 1 (post-dose) | 76795.9 (31136.7) | 74661.2 (24561.6)
  Day 3 (pre-dose): number analyzed (Participants) | 167 | 180
  Day 3 (pre-dose) | 28017.9 (11019.6) | 27738.8 (12892.4)
  Day 3 (post-dose): number analyzed (Participants) | 160 | 176
  Day 3 (post-dose) | 94653.8 (115895.1) | 87663.1 (93166.2)
  Day 17 (pre-dose): number analyzed (Participants) | 0 | 100
  Day 17 (pre-dose) |  | 4509.9 (2372.6)
  Day 17 (post-dose): number analyzed (Participants) | 0 | 153
  Day 17 (post-dose) |  | 49111.0 (71552.1)
  Day 31 (pre-dose): number analyzed (Participants) | 0 | 80
  Day 31 (pre-dose) |  | 4954.8 (4193.9)
  Day 31 (post-dose): number analyzed (Participants) | 0 | 147
  Day 31 (post-dose) |  | 67519.7 (224677.3)

10. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) to MEDI6012
Description: Number of participants with positive ADA titer to MEDI6012 are reported in 3 categories, ADA positive at any visit up to Day 70-84 follow-up visit, ADA positive with > 30% decrease in HDL-C from baseline (on the same date) at any visit up to D70-84 FU V, and ADA positive and > 30% decrease in HDL-C from baseline at Day 70-84 Follow-up Visit.
Time Frame: Predose on Day 1, Day 17, Day 31, 70 to 84 days, and on Day 195 post Day 1 dose
Population: Immunogenicity population included all treated participants, grouped according to actual treatment received and had at least one serum sample for immunogenicity testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo | Cohort A: MEDI6012 | Cohort B: Placebo | Cohort B: MEDI6012
Number analyzed (Participants) | 90 | 179 | 111 | 194
Participants
  ADA positive at any visit up to Day 70-84 Follow-up Visit | 1 | 13 | 1 | 93
  ADA positive and > 30% decrease in HDL-C from baseline at any visit up to Day 70-84 Follow-up Visit | 1 | 3 | 0 | 1
  ADA positive and > 30% decrease in HDL-C from baseline at Day 70-84 Follow-up Visit | 1 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 1 through Day 195 post Day 1 dose
Groups:
- Placebo Cohort A: Participants received placebo matched to MEDI6012 on Day 1 prior to primary percutaneous coronary intervention (pPCI) followed by a second inpatient dose on Day 3 by intravenous (IV) push.
- MEDI6012 Cohort A: Participants received loading dose of MEDI6012 300 mg on Day 1 prior to pPCI followed by a second inpatient dose of MEDI6012 150 mg on Day 3 by IV push.
- Placebo Cohort B: Participants received placebo matched to MEDI6012 on Day 1 prior to pPCI followed by a second inpatient dose on Day 3, and outpatient maintenance doses on Days 10, 17, 24, and 31 by IV push.
- MEDI6012 Cohort B: Participants received loading dose of MEDI6012 300 mg on Day 1 prior to pPCI followed by a second inpatient dose of MEDI6012 150 mg on Day 3, and outpatient maintenance doses of MEDI6012 100 mg on Days 10, 17, 24, and 31 by IV push.
Arm/Group | Placebo Cohort A | MEDI6012 Cohort A | Placebo Cohort B | MEDI6012 Cohort B
All-Cause Mortality (participants affected / at risk) | 0/90 | 2/179 | 0/111 | 1/195
Serious Adverse Events (participants affected / at risk) | 11/90 | 34/179 | 24/111 | 41/195
Other Adverse Events (participants affected / at risk) | 28/90 | 74/179 | 47/111 | 89/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cohort A (N=90) | MEDI6012 Cohort A (N=179) | Placebo Cohort B (N=111) | MEDI6012 Cohort B (N=195)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Angina unstable (Cardiac disorders) | 1 (2) | 2 (2) | 2 (3) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (3) | 5 (6) | 2 (3) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dressler's syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Torsade de pointes (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Proctitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular stent thrombosis (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis a (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin t increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatic haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post thrombotic syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cohort A (N=90) | MEDI6012 Cohort A (N=179) | Placebo Cohort B (N=111) | MEDI6012 Cohort B (N=195)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 1 (1) | 6 (6)
Angina pectoris (Cardiac disorders) | 2 (2) | 4 (5) | 4 (4) | 6 (6)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 6 (6) | 5 (5) | 7 (7)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3) | 5 (5)
Cardiac failure (Cardiac disorders) | 1 (1) | 4 (4) | 3 (4) | 9 (9)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 5 (6) | 1 (1) | 2 (2)
Supraventricular extrasystoles (Cardiac disorders) | 2 (2) | 3 (3) | 1 (1) | 3 (3)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 5 (5) | 2 (2) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2) | 8 (9)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 11 (14)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 3 (4)
Fatigue (General disorders) | 3 (3) | 4 (4) | 4 (4) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 4 (4) | 4 (4) | 3 (3)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 5 (5) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 5 (5)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 3 (3)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 2 (2) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (7) | 5 (5) | 2 (2) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 3 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (3) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 13 (13) | 5 (5) | 4 (4)
Headache (Nervous system disorders) | 4 (4) | 7 (7) | 5 (5) | 12 (13)
Anxiety (Psychiatric disorders) | 0 (0) | 4 (4) | 1 (1) | 6 (6)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 5 (5)
Renal failure (Renal and urinary disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (8) | 3 (3) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 3 (3) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Brachiocephalic arteriosclerosis (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Haematoma (Vascular disorders) | 0 (0) | 4 (4) | 2 (2) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 4 (4) | 1 (1) | 6 (6)
Hypotension (Vascular disorders) | 0 (0) | 3 (3) | 7 (7) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT03578809/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT03578809/SAP_001.pdf